CLINICAL TRIAL: NCT06411938
Title: A Community-based Cervical Cancer Prevention Program in Kenya: Overcoming Obstacles to Care, Promoting Understanding of HPV Natural History
Brief Title: A Cervical Cancer Prevention Program in Kenya
Acronym: Merck-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Academic Model Providing Access to Healthcare (AMPATH) (Other)
Responsible Party: Principal Investigator, Darron Brown MD, MPH, Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MISP 101003
Record Dates: First submitted 2024-04-03; First posted 2024-05-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer Prevention; Cervical Cancer
Keywords: Kenya; cervical cancer; prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Watchful Waiting; Acetic Acid

STUDY DESIGN:
Intervention Model Description: Community-based, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kenyan women (Other): Up to 300 adult women will undergo cervical cancer screening.
  Interventions: Diagnostic Test: High Risk HPV DNA Testing; Procedure: Visual Inspection with acetic acid (VIA) and possible cervical biopsy
- Kenyan daughters (Other): Up to 2000 girls (daughters of participants in the Kenyan women arm) will be immunized against HPV using the 9-valent HPV vaccine (Gardasil-9).
  Interventions: Biological: Gardisil-9

INTERVENTIONS:
Diagnostic Test: High Risk HPV DNA Testing — Self-collected cervical swabs will be tested for high-risk HPV using the Roche Cobas Assay. This assay provides specific HPV 16 or 18 detection, as well as detection of any of 12 additional oncogenic types (HPV types 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68).
  Arms: Kenyan women
Procedure: Visual Inspection with acetic acid (VIA) and possible cervical biopsy — Cervical screening in Kenya is usually done through pelvic examination and VIA. Cervical biopsy will additionally be performed for all HIV-infected women, and for HIV-uninfected women with abnormal VIA results.
  Arms: Kenyan women
Biological: Gardisil-9 — The 9 valent vaccine will be offered to 2000 adolescent girls. The first vaccination dose will be administered at a community meeting, after parental consent has been obtained. The second vaccination dose will be administered at a subsequent community meeting, 6 to 12 months after the first dose.
  Other Names: 9-valent HPV vaccine
  Arms: Kenyan daughters

SUMMARY:
Cervical cancer is caused by oncogenic, or "high-risk" (HR) human papillomavirus (HPV), and is the main cause of cancer-related death among Kenyan women. This malignancy is theoretically preventable through a combination of screening of adult women and treating those with cervical premalignancies and vaccination of children and adolescents against HPV infection. However, only 5% of Kenyan women are regularly screened, and only 14% have ever been screened, which in Kenya is done by a method known as Visual Inspection with Acetic Acid (VIA). Possible obstacles to current screening include long travel to clinics, high costs, poor sensitivity and specificity of VIA, the need for extensive training for VIA, variability among providers in their interpretation of VIA, lack of trained personnel, and others. In addition, while safe and effective HPV vaccines have been available for 15 years, very few (<1%) Kenyan children and adolescents have been vaccinated. Obstacles to vaccination include high costs, poor delivery infrastructure, lack of education, long travel to clinics, and others. The investigators began a community-based program in 2018 to develop a framework for eradication of cervical cancer by screening adult women and vaccinating female children. This program is becoming accepted in the Webuye region of Western Kenya, but there is still a great deal to learn.

Going forward, this initiative will be known as the Kenya Mother-Daughter Cervical Cancer Eradication Program, or the Mother-Daughter Program (MDP) for short. The investigators propose a continuation of the MDP that will allow them to accumulate additional data needed to solidify the overall project and to answer additional questions as described below. To accomplish this goal the investigators will first enroll an additional 300 adult women to the program. This will increase the strength of the analysis of HR-HPV testing in detecting premalignant lesions of the cervix, especially in HIV-infected women. Second, the investigators will identify the positive and negative features of the MDP from the viewpoint of both the adult women and the girls enrolled in the program. Third, because anogenital warts (AGWs) may serve as a reservoir for HR-HPV, especially in women living with HIV/AIDS, the investigators will examine the prevalence, HPV type distribution, and treatment of these lesions among adult women participating in the MDP.

DETAILED DESCRIPTION:
Strategies based on centralized care have been unsuccessful in preventing cervical cancer in Kenyan women. HR-HPV DNA testing of self-collected vaginal swabs is acceptable and feasible, and the investigators have now shown that such testing can occur in a community setting in rural Kenya; other groups have demonstrated similar successes in Africa. In studies funded by MISP awards, the investigators have shown that essentially all women invited to community meetings agreed to enroll in the studies, to receive education about cervical cancer, and to provide a self-collected vaginal swab for HR-HPV DNA testing. Nearly all women who attended the community meetings were also willing to have their female children vaccinated against HPV. The investigators have also shown that HPV vaccine can be delivered to western Kenya and can be administered to girls in a community setting. The investigators wish to continue to use this framework in the next MISP to further study the utility of this strategy and to address research questions that will elucidate the barriers to participation and will begin to provide information about the impact of the program.

To accomplish this goal, and an additional 300 adult women will be enrolled into the program. This will increase the strength of the proposed analysis of HR-HPV testing in detecting premalignant lesions of the cervix, especially in HIV-infected women. Second, investigators will identify the positive and negative features of the MDP from the viewpoint of both the adult women and the girls enrolled in the program. Third, because anogenital warts (AGWs) may serve as a reservoir for HR-HPV, especially in women living with HIV/AIDS, investigators will examine the prevalence, HPV type distribution, and treatment of these lesions among adult women participating in the MDP.

Thus these aims build on the infrastructure the investigators have created in the first two MISP award cycles. The investigators believe the MDP, a community based approach to cervical cancer, can become the standard for western Kenya, act as a framework for HPV-associated cancer control, and can lead to a significant improvement in patient care as well as providing an opportunity for hypothesis driven research.

ELIGIBILITY:
Kenyan Adult Women

Inclusion Criteria:

* ages 30 through 55 years
* able/willing to sign informed consent
* able to travel to Webuye clinic for VIA

Exclusion Criteria:

* unwilling to sign informed consent
* not willing or able to travel to Webuye clinic for VIA

Kenyan Girls

Inclusion Criteria:

* ages 9 through 14 years
* willing to sign informed assent for vaccination
* able to return for the second HPV vaccine dose

Exclusion Criteria:

* girls who are not willing or unable to return for the second HPV vaccine dose
* severe allergic reaction to yeast or a previous dose of the HPV vaccine

Ages: 9 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2300 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Association between biopsy-proven (CIN2/3+) VIA abnormality and HR-HPV DNA testing | Baseline
  Following a community meeting at which education on cervical cancer, self-collection of swabs for analysis and HPV vaccination are discussed, participating adult women will provide a self collected swab that will be analyzed for high risk HPV.
  All participating adult women will additionally undergo pelvic examination and VIA (the Kenyan standard of care) at a local clinic. Cervical biopsy will be performed on all women with abnormal VIA examinations, and on 10% of women who have normal VIA exams.
  Associations between biopsy-proven VIA abnormality and HR-HPV DNA status will be evaluated to obtain preliminary data for sensitivity and specificity of HR-DNA tests in the detection of biopsy-proven CIN 2/3+.
Acceptability of the Mother Daughter Program | Baseline and after HPV vaccination of daughters is complete (assessed 2 weeks after second vaccine)
  A detailed questionnaire will be used to 1) determine knowledge and beliefs of mothers about HPV and cervical cancer, which will be administered at the beginning of the study and at the end of the study, and 2) capture the opinions of mothers and daughters regarding all aspects of the program. Mothers will be asked about the self-collected swabs, travel to community meetings and the Clinic, and acceptability of HPV vaccination of daughters.
  Daughters will be asked to answer questions related to vaccination; how the community-based approach compared to a school-based program, and other questions. Children will fill out the questionnaire with help from their mothers.
  The final questionnaire will be administered two weeks after the second HPV vaccine is administered to participating daughters.

OTHER OUTCOMES:
HPV detection in genital warts | Baseline
  Genital warts will be removed and tested for HPV types

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 2 years after study completion
Access Criteria: Upon reasonable request